CLINICAL TRIAL: NCT05767931
Title: Development of Multi-specific Antibodies Based on Immune Microenvironment of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: BC-P32
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collection of biopsy specimen and surgical specimen from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, single-center, non-randomized, non-controlled study

DETAILED DESCRIPTION:
Immunotherapy with immune-checkpoint inhibitors (ICIs) has enabled a leap forward in the treatment of various types of cancer within the past decade. However,only 12.46% of patients with cancer are expected to respond to ICIs.Our team have recently developed a multi-specific antibody technology platform for the microenvironment of solid tumors.

In this study, we are going to study the tumor immune microenvironment of breast cancer patients by patient-derived organoids or PDX model，to design multi-specific antibody drugs for different tumor immune microenvironment，to look forward to improve the effectiveness of immunotherapy for breast cancer and solve the problem of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 70 years old；
2. Primary lesion >2cm on imaging examination, or suspected axillary lymph node metastasis on imaging examination；
3. Previous not received preoperative radiotherapy, chemotherapy, endocrine therapy, immunotherapy, or other anticancer treatments；
4. Subjects signed informed consent；

Exclusion Criteria:

1. A history of prior or concomitant malignancies;
2. Advanced stage breast cancer (stage IV)；
3. Suspected or confirmed lesion was surgically removed；
4. Patients were accompanied by severe organic diseases such as heart and cerebral disease, and liver and kidney disease.；

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-06 (Estimated); Primary Completion 2024-11-06 (Estimated); Study Completion 2025-03-06 (Estimated)

PRIMARY OUTCOMES:
antitumor rate of multi-specific antibody in patient-derived organoids and PDX model | 24 months
  Patient-derived organoids and PDX model

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Fan, Principal Investigator — Breast center at Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China